CLINICAL TRIAL: NCT05483881
Title: A Multicenter Observational Study of the Effects of Air Pollution on Respiratory Diseases in Children
Brief Title: the Effects of Air Pollution on Respiratory Diseases in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Tianjin Children's Hospital (Other); Jiangxi Province Children's Hospital (Other); Wuhan Children's Hospital (Other); Capital Institute of Pediatrics, China (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Guangzhou Women and Children's Medical Center (Other); The First Affiliated Hospital of Anhui Medical University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Shenzhen Children's Hospital (Other Government); Xian Children's Hospital (Other Government); The First Affiliated Hospital of Guangzhou Medical University (Other); China-Japan Friendship Hospital (Other); Kunming Children's Hospital (Other); Xianyang Children's Hospital (Other)
Responsible Party: Principal Investigator, Baoping XU, Chief of Respiratory Department Affiliation: Beijing Children's Hospital, Beijing Children's Hospital
Other Study IDs: BCH Lung 016
Record Dates: First submitted 2022-01-14; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Disease
Keywords: Respiratory Diseases; children; air pollution
MeSH Terms: conditions — Respiration Disorders; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators expect to reveal the association between air pollution and childhood respiratory diseases through a multi-center observational study, and summarize the relationship between air pollution and childhood respiratory diseases.

DETAILED DESCRIPTION:
The investigators will collect the data of outpatient and emergency children in Beijing Children's hospital and other participating hospitals due to respiratory diseases from 2010 to 2021, , collect clinical data and basic information, obtain air pollution data and meteorological monitoring data and perform data processing and statistical analysis,，then analyzes the impact of air pollution on children's respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* All children participating in this clinical study must meet all of the following criteria:

  1. Age: 0-18 years old, male and female
  2. Consultation for respiratory diseases
  3. Visit time is between 2010-2021
  4. Provide complete personally identifiable information and medical information

Exclusion Criteria:

* All children with any of the following conditions must be excluded from this study:

  1. children who visit hospital don't for respiratory diseases
  2. children participating in this clinical study don't provide complete personally identifiable information and medical information
  3. Visit time is not between 2010-2021.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children aged between 0-18 years who visited Beijing Children's hospital or other hospitals participating in the project due to respiratory diseases from 2010 to 2021.
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Major air pollutant concentrations | 12 years
  The air pollutant data comes from the daily air quality data published by the National Environmental Monitoring Center. Calculate the arithmetic average of the daily average concentrations of air pollutants (PM10, PM2.5, SO, NO, CO, etc.) Converted from air pollution index (API).

SECONDARY OUTCOMES:
Number of daily visits for respiratory diseases in outpatient and emergency departments | 12 years
  The number of daily outpatient visits for respiratory diseases( rhinitis, allergic rhinitis, upper respiratory tract infection, bronchitis and bronchiolitis, bronchiolitis obliterans, pneumonia, asthma , allergic cough, chronic cough, upper airway cough syndrome,etc.) in each hospital participating in this study during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Baoping Xu, Beijing, Beijing Municipality, China